CLINICAL TRIAL: NCT06710600
Title: Study to Assess the Photosensitizing Potential of Frequently Prescribed Medicines in Healthy Volunteers: a Pilot Study
Brief Title: Phototoxicity of Frequently Prescribed Medicines
Acronym: Phototox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Wolzt, Prof. MD, Prof., MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Phototox; 2021-000467-80 (EudraCT Number)
Record Dates: First submitted 2024-11-21; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Phototoxicity
Keywords: clinical pharmacology; phototoxicity; dermatology; adverse drug reactions
MeSH Terms: conditions — Dermatitis, Phototoxic; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): single oral dose of following medications, including 7 days wash-out phase respectively:
  1. diclofenac
  2. voriconazole
  3. hydrochlorothiazide
  4. pantoprazole
  5. amiodarone
  Interventions: Drug: Single oral dose of selected medicines, respectively; Radiation: UVA and UVB radiation
- Group 2 (Active Comparator): single oral dose of following medications, including 7 days wash-out phase respectively:
  1. acetylsalicylic acid
  2. verapamil
  3. doxycycline
  4. furosemide
  5. enalapril
  Interventions: Radiation: UVA and UVB radiation; Drug: Single oral dose of selected medicines, respectively

INTERVENTIONS:
Drug: Single oral dose of selected medicines, respectively — amiodarone (Amiodaron Arcana) 200mg, diclofenac (Diclobene) 100mg, hydrochlorothiazide (HCT G.L) 25mg, pantoprazole (Pantoloc) 40mg, voriconazole (Voriconazol Aristo®) 200mg
  Other Names: group 1
  Arms: Group 1
Radiation: UVA and UVB radiation — The skin of the inner arm will be exposed to five fixed incremental doses of UVA and UVB. Each dose will be applied to a circular area on the inner forearm of 1 cm diameter for both UVA and UVB.
Drug: Single oral dose of selected medicines, respectively — acetylsalicylic acid (ASS Genericon) 500mg, doxycycline (Doxybene) 200mg, enalapril (Enalapril "ratiopharm") 10mg, furosemide (Lasix) 40mg, verapamil (Verapabene) 80mg
  Other Names: group 2
  Arms: Group 2

SUMMARY:
This pilot trial aims to study 10 selected commonly prescribed medicines with different grade of phototoxic potential. As there is no currently established way to assess phototoxic potential in a systematic and quantitative way, we want to test a novel radiation and measurement protocol to provide more granular information for patients and providers.

DETAILED DESCRIPTION:
The purpose of this clinical study is to test ten commonly prescribed drugs with known photosensitizing properties in order to gain more detailed knowledge about the effects, which can help to make recommendations for patients who need these drugs for their therapy. Phototoxic and photoallergic drug-induced reactions are relatively common side effects of multiple drugs. However, the incidence and threshold doses are underreported, misdiagnosed or not adequately investigated.

In this open, randomized, monocentric, parallel group study, 12 healthy subjects are randomized into 2 groups of 6 healthy subjects each after fulfilling inclusion and exclusion criteria and a screening visit (demographics, medical history, laboratory parameters, vital parameters, ECG, physical examination including skin examination and baseline measurement of skin properties). In the study, one drug from a fixed block of 5 drugs allocated during randomization is administered orally as a single dose weekly (on days 1, 8, 15, 22, 29). 6 hours after drug administration, when the drugs have reached their peak plasma concentrations, the skin is irradiated with UVA, UVB and visible light at previously determined locations on the upper and lower arms and back. The irradiation is carried out using equipment that is also used in clinical routine, namely a UVA lamp from Sellamed (Germany), UVB lamps from Waldmann Medizintechnik and a slide projector for visible light radiation. In the next step, skin reactions that occur immediately after irradiation and after 24 hours are analyzed using Mexameter®, Aquaflux® and a confocal Raman microscope. In addition to the safety blood parameters, regular reserve blood samples are taken at the screening and final visits for the purpose of possible later analysis of drug levels. The subjects are asked to avoid direct sunlight for the entire duration of the study or, if this cannot be avoided, to use a high sun protection factor. The final visit (visit 12) is planned for day 36.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Male or female 18-45 years of age (limits included)
3. BMI 19-27 for males and BMI 17-25 for females
4. Vital parameters at screening within normal limits
5. Electrocardiogram without clinically significant pathologic abnormalities and with QTc values lesser than 450 ms
6. Skin type II-IV on Fitzpatrick scale (table 1)
7. Women of childbearing potential agree to use adequate birth control methods during the entire study period. For all females, negative pregnancy test at screening and once monthly is required. Acceptable methods of contraception include: oral contraceptives, intrauterine device, female or male condoms with spermicide, diaphragm with spermicide, contraceptive medication patch, contraceptive medication implant, contraceptive medication injection, abstinence, or surgical sterilization more than 3 months before randomization.

Exclusion Criteria:

1. Women known to be pregnant, lactating or having a positive or indeterminate pregnancy test
2. Lack of willingness or capacity to co-operate and comply with the study procedures appropriately
3. Failure to perform screening or baseline examinations
4. Regular use of any medication (prescription or over the counter) for prevention or treatment of any medical condition in the previous 2 months except intake of contraceptives
5. Intake of any medication throughout the active phase of the study that would interfere with the study procedure as per investigator's judgement
6. Use of dietary supplements in the previous 4 weeks, incl St. John's Wort
7. Exposure to UV-radiation (including direct or indirect sun exposure, solarium, phototherapy) or use of oral sun-protective substances and self-tanning products 2 weeks prior to first medication administration and during the entire study duration
8. Scars, previous trauma, tattoos or any other condition on the inner side of the arms that would impede the study procedures
9. Evidence of active infection requiring antibiotic therapy within 14 days prior to screening
10. Any chronic medical condition requiring chronic treatment, incl. liver disease, respiratory, cardiovascular or history of malignancies within the past two years or on current anticancer treatment
11. History of gastrointestinal pathology such as gastritis, gastric ulcers, irritable bowel disease, inflammatory bowel disease, chronic constipation
12. History of diarrhoea or emesis within the past 14 days of screening
13. History of gastrointestinal surgery with exception of appendectomy
14. History of chronic autoimmune disease incl. dermatitis requiring immunosuppressive treatment within the past two months of screening or any skin condition that induces photosensitivity
15. History of chronic skin disease potentially influencing the results (in particular skin diseases associated with photosensitivity)
16. History and/or family history of skin cancer, incl. but not limited to melanoma, basal cell carcinoma and squamous cell carcinoma.
17. Known symptomatic allergies, including food allergies or intolerances and sun allergy
18. Any clinically relevant laboratory abnormalities in screening test
19. Alcohol, cigarette or drug abuse
20. Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study
21. Presence of any condition that impacts compliance with the study procedures
22. Any underlying clinical condition that, in the opinion of the investigator, would make it very unlikely for the participant to complete the study successfully
23. Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the first study product administration, or planned use during the study period
24. Employee at the study site, spouse/partner or relative of any study staff (e.g. investigator, sub-investigators, or study nurse)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Minimal erythema dose | after 24 hours once weekly respectively, for 5 weeks in total
  To assess the Minimal Erythema Dose (MED) of 10 selected human medicines with known photosensitizing properties for UVA and UVB and the reaction to visible spectrum light 24 hours after exposure to radiation

SECONDARY OUTCOMES:
Transepidermal water loss | after 24 hours once weekly respectively, for 5 weeks in total
  To assess the transepidermal water loss (TEWL) as a marker of skin barrier function of 10 selected medicines with known photosensitizing properties 24 hours after exposure to UVA, UVB and visible spectrum light radiation.
Change in molecular skin properties | after 24 hours once weekly respectively, for 5 weeks in total
  To assess changes in skin properties on a molecular level of 10 selected medicines with known photosensitizing properties 24 hours after exposure to UVA, UVB and visible specrum light radiation
Immediate photosensitivity and phototoxicity reactions | Immediately after UV exposure once weekly, respectively, for 5 weeks in total
  To assess other immediate photosensitivity and phototoxicity reactions of 10 selected medicines with known photosensitizing properties after exposure to UVA, UVB and visible spectrum light radiation, including
  * presence of exanthema
  * presence of hyperpigmentation
  * presence of erythema
  * presence of urticaria
  * presence of pruritus
  * presence of combustion

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No